CLINICAL TRIAL: NCT06773845
Title: Building Evidence for Ablative Internal Radiation Therapy Using Yttrium-90 Glass Microspheres in Localized Hepatocellular Carcinoma Beyond the Up-To-7 Criteria
Brief Title: Building Evidence for Ablative Internal Radiation Therapy in Localized HCC Beyond the Up-To-7 Criteria
Acronym: BEAT-UT7
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Jin Woo Choi, Clinical Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2412-135-1601
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC); Radioembolization
Keywords: Hepatocellular carcinoma; Radioembolization; SIRT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radioembolization (Experimental): Ablative radioembolization using Yttrium-90 glass microspheres
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — The multicompartment MIRD model (a.k.a. partition model) based on diagnostic CT/MRI and 99mTc-MAA SPECT-CT will be used to plan a targeted dose of 700 Gy (± 50%) to the tumor. Given the high tumor burden, a scheduled second radioembolization within 120 days from the initial treatment will be permitted at the discretion of the operators provided the cumulative lung dose remains below 50 Gy. A scheduled second radioembolization may be considered when the largest tumor diameter exceeds 8 cm, or the estimated lung dose reaches 30 Gy while the tumor absorbed dose remains below the target dose of 700 Gy. The radioactive microsphere delivery device used will be glass-based (TheraSphere; Boston Scientific, MA, USA), in which Y90 is an integral constituent of the biocompatible glass matrix. Dosimetry planning will be made by personalized dosimetry software (Simplicit90y; Boston Scientific).
  Other Names: Y90 glass microsphere

SUMMARY:
At four major centers in Korea, patients with hepatocellular carcinoma (HCC) that exceed the up-to-7 criteria yet remain locally confined will undergo ablative radioembolization using Yttrium-90 glass microspheres, guided by a standardized dosimetry method. Their treatment response, survival outcomes, and adverse events will be monitored for two years following the procedure.

DETAILED DESCRIPTION:
This prospective, multi-center, open-label, single-arm, phase II clinical trial aims to evaluate the efficacy and safety of ablative radioembolization in patients with hepatocellular carcinoma (HCC) that exceeds the up-to-seven (UT7) criteria but is confined to up to five geographically adjacent Couinaud segments. The primary endpoint is the objective response rate, assessed according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST).

All patients will receive ablative radioembolization using Yttrium-90 glass microspheres with a personalized dosimetry approach targeting a tumor dose of 700 Gy (±50%). In cases of high tumor burden, a second radioembolization within 180 days of the initial procedure will be permitted at the operators' discretion, provided the cumulative lung dose remains below 50 Gy. Follow-up evaluations, including laboratory tests and dynamic imaging, will be performed at 4 weeks post-treatment and every 3 months thereafter for a total of 2 years. Efficacy data-including tumor response and survival-will be collected, with tumor responses evaluated by both site investigators and a blinded independent central review. Adverse events will be documented and graded according to the Common Terminology Criteria for Adverse Events v5.0. In addition, the incidence of radioembolization-induced liver disease and radiation pneumonitis will be monitored for 6 months following the procedure.

ELIGIBILITY:
Inclusion criteria

* Adult aged 19 and over
* HCC diagnosed by histology or non-invasive criteria of the American Association for the Study of Liver Disease
* Unresectable HCC beyond the UT7 criteria: the sum of the diameter of the largest tumor (cm) and the number of tumors > 7
* Localized HCC: all tumors are in the one to five geographically adjacent Couinaud segments
* No current or previous HCC in the untreated liver (i.e., future liver remnant [FLR])
* FLR volume > 30% of total non-tumorous liver volume
* Child-Pugh class A
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* No major organ dysfunction according to blood test performed within two months of study enrollment:

  * Leukocytes ≥ 2,000/µL and ≤ 15,000/µL
  * Hemoglobin ≥ 8.0 g/dL (transfusion allowed to meet this criterion)
  * Total bilirubin ≤ 2.0 mg/dL
  * Platelet ≥ 40,000/µL
  * International normalized ratio (INR) ≤ 2.0 for patients not taking anticoagulants
  * Aspartate transaminase (AST) ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
  * Alanine transaminase (ALT) ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
  * Creatinine ≤ 2.5 mg/dL
* Patients with a life expectancy of more than 3 months
* For women of childbearing age, a negative serum pregnancy test
* Patients who have adequately understood the clinical trial and consented in writing

Exclusion Criteria:

* HCC with vascular invasion and/or bile duct invasion on dynamic computed tomography (CT) or magnetic resonance imaging (MRI)
* HCC with extrahepatic spread on chest CT and abdominal CT or MRI
* Multinodular disseminated HCC: largest tumor size < 6 cm, or number of tumors > 10
* Patients who are not suitable for ablative radioembolization as indicated by pre-treatment mapping with 99mTc-macroaggregated albumin (MAA):

  * Cases where the estimated lung dose exceeds 30 Gy when 350 Gy of tumor absorbed dose is administered to the tumor based on the multicompartment Medical Internal Radiation Dose (MIRD) model
  * Cases with severe hepatic artery-portal vein shunting that might lead to irradiation of the non-tumorous liver segments
  * Cases where the operator determines that there is substantial adhesion with the surrounding organs such as the bowel, making ablative radioembolization infeasible
* Cases where the operator judges that the occurrence of even mild radiation pneumonitis could be fatal, based on marked emphysema or interstitial lung disease findings on chest CT
* Patients who have had active cancer within the last two years prior to the study enrollment
* History of severe allergy of intolerance to contrast agents
* Contraindication to angiography or selective visceral catheterization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to the mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with partial or complete response accroding to the mRECIST as the best response, divided by the total number of participants (%)

SECONDARY OUTCOMES:
ORR according to the RECIST 1.1 | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with partial or complete response according to the RECIST 1.1 as the best response, divided by the total number of participants (%)
ORR according to localized mRECIST and RECIST 1.1 | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with partial or complete response as the best response, divided by the total number of participants (%). In the localized mRECIST and RECIST 1.1, the tumor response is assessed only within radioembolization-treated area.
Duration of response according to mRECIST, localized mRECIST, and RECIST 1.1 | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The time from the first documentation of partial or complete response to the first occurrence of progressive disease, death from any cause, or receipt of subsequent anticancer treatment, whichever comes first.
Overall survival rate | Time of treatment up to participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Progression-free survival rates according to mRECIST, localized mRECIST, and RECIST 1.1 | Time of treatment up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time-to-progression according to mRECIST, localized mRECIST, and RECIST 1.1 | Time of treatment up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled).
Major pathologic response rate (%) after surgical resection or liver transplantation | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with major pathologic response of the largest tumor after surgical resection or liver transplantation, divided by the total number of participants who received surgical resection or liver transplanation (%). Major pathologic response refers to ≥ 90% of pathologic necrosis of the largest resected tumor
Curative conversion rate | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  Curative conversion: resection, liver transplantation, or percutaneous ablation
Sustainable complete response rate according to mRECIST more than 1 year | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Locoregional treatment unsuitability rate | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  LRT unsuitability will be determined if any of the following criteria are met.
  * Lack of objective response after two sessions of intra-arterial treatments
  * Development of new HCC within the treatment zone
  * Development of vascular invasion within the treatment zone
  * Development of extrahepatic spread
Time to and reason for subsequent HCC treatment | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Threshold tumor absorbed dose (Gy) to predict radiologic complete response and objective response as the best response by localized mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Adverse event and serious adverse event according to CTCAE v5.0 | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
The presence or absence of radiation pneumonitis diagnosed by chest simple X-ray or CT | Time of treatment up to 180 days after the initial treatment or subsequent anticancer treatment, whichever comes first
The presence or absence of radioembolization-induced liver disease | Time of treatment up to 180 days after the initial treatment or subsequent anticancer treatment, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Choi, MD, PhD, Study Chair — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - National Cancer Center, Ilsan, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No